CLINICAL TRIAL: NCT03501498
Title: The Effect of Intestinal Transit on the Entrohepatic Circulation of Bile Salts, Faecal Microbiome and Production of Volatile Organic Compounds
Brief Title: Gut Transit Effect on Enterohepatic Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16/P/138; 221556 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2021-10

CONDITIONS: Intestinal Transit
Keywords: Intestinal Transit, Bile Salts, Gut Bacteria, Volatile Organic Compounds
MeSH Terms: interventions — Loperamide; Sennosides

STUDY DESIGN:
Intervention Model Description: Randomised cross-over study. Volunteers will be assessed at baseline, then after either taking loperamide or senna at the maximally tolerated dose for 2 days prior to the 'assessment period' then during the assessment period (5-7 days). After a washout period of at least 21 days, volunteers will then repeat the same assessments but cross over to take the second drug either loperamide or senna.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- loperamide (Experimental): Slows intestinal transit time
  Interventions: Drug: Loperamide
- senna (Experimental): Speeds up intestinal transit time
  Interventions: Drug: Senna

INTERVENTIONS:
Drug: Loperamide — Alters intestinal transit time.
  Arms: loperamide
Drug: Senna — Alters intestinal transit time.
  Arms: senna

SUMMARY:
A study to determine the influence of changing intestinal transit time of the enterohepatic recirculation of bile acids.

DETAILED DESCRIPTION:
The digestion of food by human body starts from oral cavity and continues until its excreted as faeces. There are different factors affecting this process. Important factors are movement through the GI Tract, breakdown of food material and absorption by the body to produce energy. The unabsorbed waste material is then excreted by the body.

Different enzymes are produced by human body which are responsible for digestion of food. One important chemical is bile which is produced in the gall bladder. It is important in digestion of fatty foods but affects the movement of food material as well. There are numerous bacteria present in human GI tract especially in mouth and large bowel which also play an important role in process of digestion of food.

Different conditions of health and disease can affect how food moves through the GI tract (known as intestinal transit). It also affects the activity of different digestive enzymes and chemicals in body. The bacterial population in the body is also affected by changes described above. The purpose of this study is to observe how these different processes especially the intestinal transit, bile salts and gut bacteria affect each other. This will help to identify mechanisms responsible for different disorders of human gut like irritable bowel syndrome. The study is part of an effort to identify new and future treatment of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy volunteers between the ages of 18 and 65

Exclusion Criteria:

* Unable to consent
* Pregnant or lactating
* Known diarrhoeal disorder
* Known constipation.
* Any gastrointestinal disease or previous gastric surgery
* An episode of gastroenteritis within the last month
* Taking any acid suppressing medication
* Any significant medical condition (e.g. diabetes, renal disease)
* Any antibiotic intake within the last one-month
* Any drug with known effects on GI motility
* Known allergy or intolerance to senna or loperamide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The effect of intestinal transit on faecal bile acids | 7 days
  Change in bile acid pool and activity from baseline with each intervention

SECONDARY OUTCOMES:
Stool bacterial count | 7 days
  Bacterial count
1. common stool test | 7 days
  calprotectin
2. common stool test | 7 days
  elastase
3. common stool test | 7 days
  lactoferrin
Volatile Organic Compounds | 5 days
  VOC estimation in urine

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lewis, MD, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Derriford Hospital, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No